CLINICAL TRIAL: NCT00664027
Title: An Open-Label, Randomized, Dose-ranging Phase IIa Trial to Determine the Effects of RTA 402 (Bardoxolone Methyl) on Renal Function in Patients With Diabetic Nephropathy
Brief Title: Phase IIa Trial to Determine the Effects of Bardoxolone Methyl on Renal Function in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTA 402-C-0801
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — bardoxolone methyl

ARMS (4):
- 25 mg (Experimental): 25 mg RTA 402 (Bardoxolone methyl)/Stratum 1
  Interventions: Drug: RTA 402 (Bardoxolone Methyl)
- 75 mg (Experimental): 75 mg RTA 402 (Bardoxolone methyl)/Stratum 1
  Interventions: Drug: RTA 402 (Bardoxolone Methyl)
- 150 mg (Experimental): 150 mg RTA 402 (Bardoxolone methyl)/Stratum 1
  Interventions: Drug: RTA 402 (Bardoxolone Methyl)
- 25/75 mg (Experimental): 25 mg -> 75 mg RTA 402 (Bardoxolone methyl)/Stratum 2
  Interventions: Drug: RTA 402 (Bardoxolone Methyl)

INTERVENTIONS:
Drug: RTA 402 (Bardoxolone Methyl) — Stratum 1: 25, 75, 150mg/day, orally, 28 consecutive days Stratum 2: 25 mg/day, orally, 28 consecutive days followed by 75 mg/day, orally, 28 consecutive days

SUMMARY:
To determine the effects of three different doses of bardoxolone methyl administered orally on the kidney function (glomular filtration rate) in patients with diabetic nephropathy.

DETAILED DESCRIPTION:
Bardoxolone methyl is an Antioxidant Inflammation Modulator in clinical development for inflammation and cancer-related indications that inhibits immune-mediated inflammation by restoring redox homeostasis in inflamed tissues. It induces the cytoprotective transcription factor Nrf2 and suppresses the activities of the pro-oxidant and pro-inflammatory transcription factors NF-kB and the STATs. In vivo, bardoxolone has demonstrated significant single agent anti-inflammatory activity in several animal models of inflammation such as renal damage in the cisplatin model and ischemia-reperfusion model of acute renal injury. In addition, significant reductions in serum creatinine have been observed in patients treated with bardoxolone. Based on these data, it is hypothesized that bardoxolone can improve renal function in patients with diabetic nephropathy through suppression of renal inflammation and improvement of glomerular filtration.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes;
2. Serum creatinine in women 1.3 - 3.0 mg/dL (115-265 μmol/L), inclusive, and in men 1.5 - 3.0 mg/dL (133-265 μmol/L), inclusive;
3. Patient must agree to practice effective contraception.
4. Patient must have a negative urine pregnancy test within 72 hours prior to the first dose of study medication.
5. Patient is willing and able to cooperate with all aspects of the protocol and is able to communicate effectively.
6. Patient is willing and able to provide written informed consent to participate in this clinical study.

Exclusion Criteria:

1. Type 1 (insulin-dependent; juvenile onset) diabetes.
2. Patients with known non-diabetic renal disease (nephrosclerosis superimposed on diabetic nephropathy acceptable), or with renal allograft.
3. Cardiovascular disease as follows: unstable angina pectoris within 3 mo of study entry; myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 3 mo of study entry; transient ischemic attack within 3 mo of study entry; cerebrovascular accident within 3 mo of study entry; obstructive valvular heart disease or hypertrophic cardiomyopathy; second or third degree atrioventricular block not successfully treated with a pacemaker.
4. Need for chronic (>2 weeks) immunosuppressive therapy, including corticosteroids (excluding inhaled or nasal steroids) within 3 mo of study entry.
5. Evidence of hepatic dysfunction including total bilirubin >1.5 mg/dL (>26 micromole/L); elevation of liver transaminase (aspartate aminotransferase [AST] or alanine transferase [ALT])above the upper limit of normal(ULN) within the 14-day screening period; documented elevation (above ULN) of AST or ALT within 3 months prior to screening; elevation of alkaline phosphatase (ALP) above 1.5 x ULN; documented elevation of gamma-glutamyl transpeptidase (GGT) above 1.5 X ULN.
6. If female, patient is pregnant, nursing or planning a pregnancy.
7. Patient has any concurrent clinical conditions that in the judgment of the investigator could either potentially pose a health risk to the patient while involved in the study or could potentially influence the study outcome;
8. Patient has known hypersensitivity to any component of the study drug;
9. Patient has known allergy to iodine;
10. Patient has undergone diagnostic or intervention procedure requiring a contrast agent within the last 30 days prior to entry into the study;
11. Change or dose-adjustment in any of the following medications: ACE inhibitors, angiotensin II blockers, non-steroidal anti inflammatory drugs (NSAIDs), or COX-2 inhibitors within 3 months; other anti-hypertensive, and other anti-diabetic medications within 6 weeks prior to entry into the study;
12. Patient has a history of drug or alcohol abuse or has positive test results for any drug of abuse (positive urine drug test and/or alcohol breathalyzer test).
13. Patients who are unable or unwilling to discontinue the following medications until 1 week following last dose of study treatment: Nicotinic acid, Isoniazid, Dantrolene, Labetalol, Pemoline, Felbamate, Zileutan, Tolcapone, Trovafloxacin, Vitamin D, Vitamin D analogues (such as Calcitriol, paricalcitol, doxercalciferol), or multivitamins containing vitamin D or related analogs, or Fenofibrate. Patient must have been off the aforementioned medications for a minimum of two weeks prior to enrollment.
14. Patient with an intact parathyroid hormone (iPTH) level > 300 pg/mL.
15. Patient has participated in another clinical study involving investigational or marketed products within 30 days prior to entry into the study or would concomitantly participate in such a study.
16. Patient is unable to communicate or cooperate with the Investigator due to language problems, poor mental development or impaired cerebral function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04-30 (Actual); Primary Completion 2009-05-31 (Actual); Study Completion 2009-05-31 (Actual)

PRIMARY OUTCOMES:
To determine the effects of RTA 402 administered orally at three dose strengths on the glomerular filtration rate (as estimated by the MDRD formula) in patients with diabetic nephropathy (stratum 1). | 28 days
To determine the effects of RTA 402 on glomerular filtration rate (as estimated by the MDRD formula) when administered for 28 days at dose of 25 mg followed by a dose of 75 mg for another 28 days in patients with diabetic nephropathy (stratum 2). | 56 days

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of oral RTA 402 administered orally at three dose strengths in patients with diabetic nephropathy. | 28 days
To evaluate the effects of RTA 402 on the serum creatinine level, iohexol serum clearance (one study center only), creatinine clearance, and urine albumin/creatinine ratio in patients with diabetic nephropathy. | 28 days (stratum 1), 56 days (stratum 2)
To evaluate the effects of RTA 402 on hemoglobin A1c in all patients enrolled and on insulin response by the hyperinsulinemic euglycemic clamp test in patients enrolled at only one of the study centers. | 28 days (stratum 1), 56 days (stratum 2)
To evaluate the effects of RTA 402 on a panel of markers of inflammation, renal injury, oxidative stress, and endothelial cell dysfunction. | 28 days (stratum 1), 56 days (stratum 2)
To determine the safety and tolerability of RTA 402 when the dose is escalated after 28 days in patients with diabetic nephropathy from 25 mg to 75 mg and continued for another 28 consecutive days. | 28 days (stratum 1), 56 days (stratum 2)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - West Houston Clinical Research Services, Houston, Texas
  - Renal Associates, PA, San Antonio, Texas
  - DGD Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/